CLINICAL TRIAL: NCT02002247
Title: SodiUm SeleniTe Adminstration IN Cardiac Surgery (SUSTAIN CSX®-Trial). A Multicentre Randomized Controlled Trial of High Dose Sodium-selenite Administration in High Risk Cardiac Surgical Patients
Brief Title: SodiUm SeleniTe Adminstration IN Cardiac Surgery (SUSTAIN CSX®-Trial).
Acronym: SUSTAINCSX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daren K. Heyland (Other)
Collaborators: biosyn Arzneimittel GmbH (Industry); Queen's University (Other); RWTH Aachen University (Other)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Scientific Director, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUSTAIN CSX
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Heart Disease
Keywords: antioxidants; selenium; heart disease; cardiac surgery; perioperative
MeSH Terms: conditions — Heart Diseases | interventions — Sodium Selenite; Selenium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Normal saline will be administered to subjects intravenously pre-operatively, upon admission to the ICU, then daily up to post-operative day 10 or ICU discharge, whichever occurs first.
  Interventions: Drug: Placebo
- sodium selenite (Active Comparator): High-dose sodium-selenite will be administered to subjects intravenously:
  1) pre-operatively (2000 ug); 2) upon admission to the ICU (2000 ug), 3) then daily (1000 ug) up to post-operative day 10 or ICU discharge, whichever occurs first.
  Interventions: Drug: sodium selenite

INTERVENTIONS:
Drug: sodium selenite — All subjects will receive an IV bolus of 2000µg selenium within 30min after induction of anesthesia via the central venous catheter. After termination of surgery, immediately after admission to the ICU, all patients will receive a second bolus of 2000µg selenium. Then on every further morning during ICU-stay, patients will receive an IV bolus of 1000µg selenium via central or peripheral venous access until death, discharge from ICU to the ward, or for a maximum of 10 days.
  Other Names: selenium
  Arms: sodium selenite
Drug: Placebo — All patients will receive an IV bolus of normal saline (equals to 40ml prepared solution) within 30min after induction of anesthesia via the central venous catheter. After termination of surgery, immediately after admission to the ICU, all patients will receive a second bolus of normal saline accordingly. Then on every further morning during ICU-stay, patients will receive an IV bolus of normal saline via central or peripheral venous access until death, discharge from ICU to the ward (treatment may continue in a step down or intermediate care unit), or for a maximum of 10 days.
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
The aim of the investigators' research program is to investigate the effects of perioperative high dose selenium supplementation in high-risk cardiac surgical patients undergoing complicated open heart surgery. The investigators hypothesize that the therapeutic strategy tested in this randomized trial may contribute to a fewer complications, less organ injury and fewer deaths. Before the investigators conducted the large definitive trial, they conducted a pilot study to assess the feasibility of the protocol, and are rolling the pilot patients into the definitive trial.

DETAILED DESCRIPTION:
Over a million patients undergo open heart surgery annually and this number is likely to accelerate as the population ages and the prevalence of diabetes and cardiovascular disease continue to increase. Unfortunately, death, organ failure, and other serious complications are all too frequent following open heart surgery, especially in some high-risk patient populations.

Selenium is a trace element that is important for many of the body's regulatory and metabolic functions especially during times of stress. International members of the study team have shown in a non-randomized study that high dose selenium supplementation was associated with improved clinical outcomes compared to a historical control group. The next step in this program of research is to conduct a randomized trial.

The aim of this research program is to investigate the effects of perioperative high dose selenium supplementation in high-risk cardiac surgical patients undergoing complicated open heart surgery. The investigators hypothesize that the therapeutic strategy tested in this randomized trial may contribute to fewer complications, less organ injury and fewer deaths.

The investigators propose to conduct a randomized, placebo-controlled, double-blind, multicentre definitive trial of 1400 patients across 20 sites in Germany and Canada, which will include the pilot study patients. An industry partner (Biosyn) will provide the product and some additional support for the European sites. Patients will be randomized to receive either a daily perioperative high-dose selenium or placebo until postoperative day 10 (maximum) or upon earlier discharge from ICU. If the hypothesis is proven true, and this simple, inexpensive nutrient reduces complications and improves recovery of patients undergoing cardiac surgery, there is the potential to dramatically change clinical practice and improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>/=18 years of age)
* Scheduled to undergo elective or urgent cardiac surgery with the use of cardiopulmonary bypass (CPB) and cardioplegic arrest that exhibit a high perioperative risk profile as defined by the presence of one or more of the following:

  * a) Planned valve surgery combined with CABG or multiple valve replacement/repair surgeries or combined cardiac surgical procedures involving the thoracic aorta; OR
  * b) Any cardiac surgery with a high perioperative risk profile, defined as a predicted operative mortality of ≥ 5% (EuroSCORE II).

Exclusion Criteria:

We will exclude patients who meet any of the following criteria:

* Isolated procedures (CABG only or valve)
* Known hypersensitivity to sodium-selenite or to any of the constituents of the solution.
* Renal failure requiring dialysis at the point of screening.
* Chronic liver disease as evidenced by a pre-operative total bilirubin >2 mg/dl or 34 umol/L.
* Disabling neuropsychiatric disorders (severe dementia, severe Alzheimer's disease, advanced Parkinson's disease).
* Pregnancy or lactation period.
* Simultaneous participation in another clinical trial of an experimental therapy (co-enrolment acceptable in observational studies or randomized trials of existing therapies if permitted by both steering committees and local ethics boards).
* Patients undergoing heart transplantation or preoperative planned LVAD insertion or complex congenital heart surgery.
* Alternate contacts of investigators (required by German Regulatory Authorities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-02 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
PODS free days + alive | 30 Day
  Evaluate the PODS free days + alive as the primary outcome for the large-scale Phase III trial. We define PODS as the need for life-sustaining therapies (mechanical ventilation, vasopressor therapy, mechanical circulatory support, continuous renal replacement therapy, or intermittent hemodialysis).

SECONDARY OUTCOMES:
30-Day Mortality | 30 Day
  Mortality 30 days post-randomization.
Hospital Acquired Infections | 30 day
  To be evaluated up to 6 months post-randomization.
Perioperative hemodynamic profile | 6 months
  This includes: mean arterial blood pressure, cardiac power index, systemic vascular resistance, etc... To be assessed up to 6-months post-randomization.
Cardiovascular Complications | 6-months
  This includes: arrhythmias, cardiac arrest, infarction. To be assessed up to 6-months.
Duration of Mechanical Ventilation | 6-months
  To be assessed up to 6-months.
Incidence of post-operative delirium | 6-months
  Assessed by CAM-ICU score. To be assessed up to 6-months.
ICU Length of stay | 6-months
  To be assessed up to 6 months post-randomization.
Hospital Re-admission Rates | 6-months
  To be assessed up to 6-months post-randomization.
Hospital Length of stay | 6-months
  To be assessed up to 6 months post-randomization.
6-Month Survival | 6-months
  To be assessed at 6 months post-randomization.
Quality of Life | 6-months
  Health related quality of life to be assessed up to 6-months post-randomization.
Return to work | 6-months
  Assessed using a questionnaire to determine the patient's ability to return to their pre-operative working capabilities. To be assessed up to 6 months post-randomization.
6-minute walking test | up to 3 months
  6-minute walking distance

OTHER OUTCOMES:
Laboratory outcomes | POD 10
  To be assessed up to post-operative day (POD) 10 in patients who consent to this optional blood work.
  To assess the potential effects of supplementation on selenium levels, safety parameters and other mechanistic markers. Whole blood levels of selenium, selenoprotein P (Sel-P), antibodies against oxidized LDL, markers of inflammation (interleukin[IL]-6, IL-10, TNF alpha) and activity of glutathione-peroxidase (GPx) will be assessed to determine the efficacy of selenium supplementation in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Queen's University; Christian Stoppe, MD, Principal Investigator — RWTH Aachen University Hospital; Bernard J McDonald, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (23):
- Canada (12):
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Institut de cardiologie de Montreal, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Sacre Coeur, Montreal, Quebec
  - IUCPQ, Québec, Quebec
  - Centre de recherche CIUSSS de l'Estrie CHUS, Sherbrooke, Quebec
- Germany (11):
  - RWTH Aachen University Hospital, Aachen
  - Klinik und Poliklinik für Anästhesiologie und Operative Intensivmedizin Universitätsklinikum Bonn, Bonn
  - Klinik und Poliklinik für Herz- und Thoraxchirurgie Uniklinik Köln, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinik für Her- und Gefäßchirurgie Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Klinik für Herz-, Kinderherz- und Gefäßchirurgie UKGM Giessen, Giessen
  - University Medical Center Schleswig-Holstein, Kiel
  - Klinik für Anästhesiologie Universitätsmedizin Mainz, Mainz
  - Klinik für Anästhesiologie Klinikum der Universität München, München
  - Klinik für Anästhesiologie, operative Intensivmedizin und Schmerztherapie Universitätsmedizin Münster, Zentralklinikum, Münster
  - Klinikum Oldenburg gGmbH Universitätsklinik für Anästhesiologie / Intensivmedizin / Notfallmedizin / Schmerztherapie, Oldenburg

REFERENCES:
- [Derived] Stoppe C, McDonald B, Meybohm P, Christopher KB, Fremes S, Whitlock R, Mohammadi S, Kalavrouziotis D, Elke G, Rossaint R, Helmer P, Zacharowski K, Gunther U, Parotto M, Niemann B, Boning A, Mazer CD, Jones PM, Ferner M, Lamarche Y, Lamontagne F, Liakopoulos OJ, Cameron M, Muller M, Zarbock A, Wittmann M, Goetzenich A, Kilger E, Schomburg L, Day AG, Heyland DK; SUSTAIN CSX Study Collaborators. Effect of High-Dose Selenium on Postoperative Organ Dysfunction and Mortality in Cardiac Surgery Patients: The SUSTAIN CSX Randomized Clinical Trial. JAMA Surg. 2023 Mar 1;158(3):235-244. doi: 10.1001/jamasurg.2022.6855. PMID 36630120
- [Derived] Stoppe C, McDonald B, Rex S, Manzanares W, Whitlock R, Fremes S, Fowler R, Lamarche Y, Meybohm P, Haberthur C, Rossaint R, Goetzenich A, Elke G, Day A, Heyland DK. SodiUm SeleniTe Adminstration IN Cardiac Surgery (SUSTAIN CSX-trial): study design of an international multicenter randomized double-blinded controlled trial of high dose sodium-selenite administration in high-risk cardiac surgical patients. Trials. 2014 Aug 28;15:339. doi: 10.1186/1745-6215-15-339. PMID 25169040

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT02002247/SAP_000.pdf